CLINICAL TRIAL: NCT01763840
Title: Contrast Enhanced Ultrasound for Evaluation of Pediatric Abdominal Trauma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: David Mooney (Other)
Responsible Party: Sponsor-Investigator, David Mooney, Associate Professor of Surgery, Boston Children's Hospital
Organization: Boston Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P00004754
Record Dates: First submitted 2013-01-04; First posted 2013-01-09 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Abdominal Trauma
Keywords: Pediatric Abdominal Trauma Ultrasound Contrast
MeSH Terms: conditions — Abdominal Injuries | interventions — FS 069

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Contrast enhanced Ultrasound (Experimental): Presence and grade of solid organ injury on contrast enhanced ultrasound
  Interventions: Drug: Contrast enhanced Ultrasound

INTERVENTIONS:
Drug: Contrast enhanced Ultrasound — Ultrasound, then contrast enhanced ultrasound.
  Other Names: Optison

SUMMARY:
The research protocol aims to compare the utility of contrast enhanced abdominal sonography with computerized tomography in the evaluation of children with blunt abdominal trauma. Hemodynamically stable children ages 7-18 who are transferred to Children's Hospital on the trauma service with a CT scan of abdomen & pelvis already performed at the referring institution will be identified by the trauma service as eligible for inclusion.

The ultrasounds will be performed by one of two Attending Radiologists involved in the study. The contrast being used for the study is Optison (GE Healthcare Inc, Princeton, NJ), which is an injectable suspension of Perflutren Protein-Type A Microspheres. This has been used in echocardiography as well as abdominal ultrasonography for evaluation of pediatric abdominal and pelvic solid tumors. The contrast enhanced ultrasound will be performed by radiologist. Contrast enhancement only lasts for 3-5 minutes per injection, therefore Optison will be redosed up to 2 additional doses for the completion of the ultrasound. Vital signs will be monitored for 30 minutes after the contrast agent is given and any adverse reactions will be recorded. Adverse reactions to Optison have occurred within this time frame in the literature. Subsequent medical care will be as indicated per the clinical practice guideline.

DETAILED DESCRIPTION:
Contrast enhanced ultrasound has been used clinically in Europe for the past 10 years as an evaulation tool for examining abdominal injuries in trauma among children and adults. This is a valuable diagnostic modality that could potentially reduce the need for radiation exposure from abdominal computed tomography (CT) scans in trauma evaluation. The research protocol aims to compare the utility of contrast enhanced abdominal sonography with computerized tomography in the evaluation of children with blunt abdominal trauma. Hemodynamically stable children ages 7-18 who are transferred to Children's Hospital on the trauma service with a CT scan of abdomen & pelvis already performed at the referring institution will be identified by the trauma service as eligible for inclusion. Children who are hemodynamically unstable, known cardiac abnormality, unable to roll over, or unable to assent will be excluded from the study. If the child is enrolled in the study, he/she will have a non contrast ultrasound, followed by a contrast enhanced ultrasound performed in the Radiology Department once he/she is stabilized and evaluation is completed in the Emergency Room. The patient will have vital signs (including blood pressure, heart rate, respiratory rate, oxygen saturation) monitored during the study and 30 minutes after contrast administration.

The ultrasounds will be performed by one of two Attending Radiologists involved in the study. The contrast being used for the study is Optison (GE Healthcare Inc, Princeton, NJ), which is an injectable suspension of Perflutren Protein-Type A Microspheres. This has been used in echocardiography as well as abdominal ultrasonography for evaluation of pediatric abdominal and pelvic solid tumors. After the non contrast ultrasound is performed, the Optison contrast agent will be given via peripheral IV. The contrast enhanced ultrasound will be performed by radiologist. Contrast enhancement only lasts for 3-5 minutes per injection, therefore Optison will be redosed up to 2 additional doses for the completion of the ultrasound. Vital signs will be monitored for 30 minutes after the contrast agent is given and any adverse reactions will be recorded. Adverse reactions to Optison have occurred within this time frame in the literature. Subsequent medical care will be as indicated per the clinical practice guideline.

ELIGIBILITY:
Inclusion Criteria:

* Hemodynamically stable
* Age 10-18 years
* Transferred to BCH Emergency Department to the Trauma Service for evaluation and management
* Concern for blunt abdominal injury
* CT A/P performed at referring institution
* Planned for admission to the hospital on the trauma service

Exclusion Criteria:

* Patients who are hemodynamically unstable
* Known cardiac abnormality
* Pulmonary hypertension
* Known sensitivity to human albumin or blood products
* Unable to roll over
* Unable to assent
* Pregnant
* Lactating

Ages: 2 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2013-04; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Primary outcome measured will be the identification of intra-abdominal injury | Baseline

SECONDARY OUTCOMES:
Secondary outcome will be assessment of grade of solid organ injury. | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jill Zalieckas, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Dolan MS, Gala SS, Dodla S, Abdelmoneim SS, Xie F, Cloutier D, Bierig M, Mulvagh SL, Porter TR, Labovitz AJ. Safety and efficacy of commercially available ultrasound contrast agents for rest and stress echocardiography a multicenter experience. J Am Coll Cardiol. 2009 Jan 6;53(1):32-8. doi: 10.1016/j.jacc.2008.08.066. PMID 19118722
- [Background] Abdelmoneim SS, Bernier M, Scott CG, Dhoble A, Ness SA, Hagen ME, Moir S, McCully RB, Pellikka PA, Mulvagh SL. Safety of contrast agent use during stress echocardiography in patients with elevated right ventricular systolic pressure: a cohort study. Circ Cardiovasc Imaging. 2010 May;3(3):240-8. doi: 10.1161/CIRCIMAGING.109.895029. Epub 2010 Mar 16. PMID 20233859
- [Background] Darge K; CEUS task force of the Society for Pediatric Radiology. Contrast-enhanced US (CEUS) in children: ready for prime time in the United States. Pediatr Radiol. 2011 Nov;41(11):1486-8. doi: 10.1007/s00247-011-2240-y. Epub 2011 Sep 22. No abstract available. PMID 21938505
- [Background] McCarville MB. Contrast-enhanced sonography in pediatrics. Pediatr Radiol. 2011 May;41 Suppl 1:S238-42. doi: 10.1007/s00247-011-2005-7. Epub 2011 Apr 27. PMID 21523607
- [Background] McCarville MB, Kaste SC, Hoffer FA, Khan RB, Walton RC, Alpert BS, Furman WL, Li C, Xiong X. Contrast-enhanced sonography of malignant pediatric abdominal and pelvic solid tumors: preliminary safety and feasibility data. Pediatr Radiol. 2012 Jul;42(7):824-33. doi: 10.1007/s00247-011-2338-2. Epub 2012 Jan 17. PMID 22249601
- [Background] McMahon CJ, Ayres NA, Bezold LI, Lewin MB, Alonzo M, Altman CA, Kovalchin JP, Eidem BW, Pignatelli RH. Safety and efficacy of intravenous contrast imaging in pediatric echocardiography. Pediatr Cardiol. 2005 Jul-Aug;26(4):413-7. doi: 10.1007/s00246-004-0795-1. PMID 16374692
- [Background] Valentino M, Serra C, Pavlica P, Labate AM, Lima M, Baroncini S, Barozzi L. Blunt abdominal trauma: diagnostic performance of contrast-enhanced US in children--initial experience. Radiology. 2008 Mar;246(3):903-9. doi: 10.1148/radiol.2463070652. Epub 2008 Jan 14. PMID 18195385
- [Background] Wei K, Mulvagh SL, Carson L, Davidoff R, Gabriel R, Grimm RA, Wilson S, Fane L, Herzog CA, Zoghbi WA, Taylor R, Farrar M, Chaudhry FA, Porter TR, Irani W, Lang RM. The safety of deFinity and Optison for ultrasound image enhancement: a retrospective analysis of 78,383 administered contrast doses. J Am Soc Echocardiogr. 2008 Nov;21(11):1202-6. doi: 10.1016/j.echo.2008.07.019. Epub 2008 Oct 10. PMID 18848430